CLINICAL TRIAL: NCT06035783
Title: Calcium Reduction by Orbital Atherectomy in Western Europe
Acronym: CROWN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Wijnand den Dekker, Interventional Cardiologist, Erasmus Medical Center
Other Study IDs: NL81318.078.22
Record Dates: First submitted 2023-03-10; First posted 2023-09-13 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2023-09

CONDITIONS: Vascular Calcification* / Diagnostic Imaging; Atherectomies, Coronary; Tomography, Optical Coherence; Coronary Intervention, Percutaneous; Coronary Angiography; Humans; Treatment Outcome; Vascular Calcification* / Therapy; Vascular Calcification
MeSH Terms: conditions — Vascular Calcification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Observational cohort: Patients undergoing PCI of a severely calcified coronary lesion in need of OA to enable proper stent placement
  Interventions: Device: Orbital Atherectomy

INTERVENTIONS:
Device: Orbital Atherectomy — The Diamondback 360° Coronary orbital atherectomy system (OAS) is a device dedicated to debulk severely calcified coronary lesions to facilitate stent delivery and enable stent expansion with optimal results. The OAS's main mechanism is the synergistic rotation of the crown around its axis and simultaneously its endoluminal orbital motion. This effect allows blood to flow continuously and it facilitates heat dispersion which results in reduced heat damage to the arterial walls and subsequently to less myocardial damage, at the same time it softens the plaques tissue. It also appears that the microparticles created from sanding the artery plaques do not create any agglomeration to the branching arteries
  Other Names: DIAMONDBACK 360 CORONARY ORBITAL ATHERECTOMY SYSTEM

SUMMARY:
In calcified lesions, optimal stent placement and expansion may prove to be challenging. Lesion preparation is necessary to facilitate optimal stenting in calcified lesions, for which orbital atherectomy can used. Therefore the aim of this study is to:

1. Show that orbital atherectomy effectuates optimal stent expansion
2. Investigate the mechanics of lesion preparation when using orbital atherectomy

Patients presenting with a significant and severely calcified lesion in need of orbital atherectomy will undergo optical coherence tomography guided orbital atherectomy and stent placement.

DETAILED DESCRIPTION:
The Diamondback 360° Coronary Orbital Atherectomy System (OAS) (Cardiovascular Systems Inc., St. Paul,MN,USA) is a percutaneous device indicated to modify calcified lesion in order to facilitate stent delivery in patients with severely calcified coronary artery disease (CAD). As of to date, detailed sequential intravascular imaging data unraveling the exact calcium modifying effect of orbital atherectomy (OA) prior to stent placement in vivo, are lacking.

The aim of this, international, multicenter, prospective and observational single arm study is to understand the mechanism of action of OA for the treatment of de novo, severely calcified coronary lesions priot to stent placement using optical coherence tomography (OCT) and to assess stent expansion, based on OCT derived minimal stent area. The study population consists of patients undergoing percutaneous coronary intervention of a severely calcified coronary lesion in need of OA to enable proper stent placement and expansion.

A total of 100 patients will be enrolled. All patients will undergo peri-procedural imaging using OCT and the aim is to obtain data for at least 50 patients with OCT before and after OA and after stenting.

ELIGIBILITY:
Inclusion Criteria:

* De novo significant native coronary artery lesion
* The target lesion must have evidence of severe calcification: 1) presence of radiopacities noted without cardiac motion prior to contrast injection involving both sides of the arterial wall with calcification length of at least 15 mm and extend partially into the target lesion. 2) OR presence of ≥ 270° of calcium or lumen protruding calcified nodules at >1 cross section by intravascular imaging (OCT)
* The target vessel reference diameter ≥ 2.5 mm and ≤ 4.0 mm and lesion must not exceed 40 mm in length

Exclusion Criteria:

* Left main disease
* Prior stenting of the target vessel
* Target lesion has thrombus or dissection
* Known left ventricular ejection fraction LVEF ≤ 25%
* Diagnosed with chronic renal failure (GFR < 30 ml/min)
* Confirmed pregnancy
* Life expectancy < 12 months
* Coronary anatomy that prevents delivery of OCT catheter
* Known allergy to soybean oil, egg yolk phospholipids, glycerin or sodium hydroxide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing PCI of severely calcified coronary lesion in need of orbital atherectomy to enable proper stent placement and expansion
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Primary imaging endpoint | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Proportion of patients that reach stent expansion ≥ 5.5mm² as assessed by OCT derived MSA

SECONDARY OUTCOMES:
Procedural success | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  Procedural success is defined as successful stent delivery with:
  1. Final core lab defined TIMI III flow
  2. Angiographic in-stent DS ≤20%
  3. absence of in-hospital major adverse cardiac and cerebrovascular events (consisting of all-cause death, spontaneous myocardial infarction, target vessel revascularization or stroke)
Target vessel failure (TVF) | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours, 30 days, 12 months
  TVF is defined as a composite of cardiac death, target vessel spontaneous myocardial infarction and target vessel revascularization.
Major adverse cardiac events (MACE) | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours, 30 days, 12 months
  MACE is defined is a composite of all-cause death, spontaneous myocardial infarction and repeat revascularization
Individual components of MACE and TVF | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours, 30 days, 12 months
  The components of MACE and TVF will be measured individually, namely:
  * All-cause death
  * Cardiac death
  * Spontaneous myocardial infarction
  * Target vessel spontaneous myocardial infarction
  * Target vessel revascularization
  * Repeat revascularization
Periprocedural myocardial infarction | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours
  The incidence of periprocedural myocardial infarction, namely type 4a (4th universal definition of myocardial infarction)
Major intraprocedural complications | Periprocedure
  Major intraprocedural complications include type C-F dissections, perforations, slow flow or no reflow, thrombus and major side branch occlusion (> 2mm)
Probable and definite stent thrombosis | Time of PCI Procedure - participants will be followed for the duration of hospital stay, an expected average of 24 hours, 30 days, 12 months
MSA on OCT | Periprocedure
  Final MSA
Stent expansion on OCT | Periprocedure
  Percentage of stent expansion
Intracoronary imaging endpoints on OCT | Periprocedure
  Minimal lumen area post orbital atherectomy and post stenting
Calcium and fractures on OCT | Periprocedure
  * Number of calcium fractures
  * Number of calcium factures based on calcium thickness post orbital atherectomy
  * Number of calcified nodules modified post orbital atherectomy
Hematoma on OCT | Periprocedure
  * Incidence of OCT defined hematomas post orbital atherectomy
  * Incidence and quantifications of dissections post orbital atherectomy
Diameter stenosis on angiography | Periprocedure
  - In-stent and in-segment DS
minimal luminal diameter Diameter on angiography | Periprocedure
  - In-stent and in-segment MLD
Acute gain Diameter on angiography | Periprocedure
  - In-stent and in-segment acute gain

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands